CLINICAL TRIAL: NCT06199921
Title: Atorvastatin-containing Treatment Regimens for Pulmonary Tuberculosis: A Randomized, Open-label, Controlled phase2C/3 Clinical Trial
Brief Title: ATORvastatin in Pulmonary TUBerculosis
Acronym: ATORTUB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Open Philanthropy (Other)
Responsible Party: Principal Investigator, Adewole Olufemi, Professor, Obafemi Awolowo University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC/2023/11/15; IRB/IEC/0004553 (Other: International)
Record Dates: First submitted 2023-12-03; First posted 2024-01-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Tuberculosis; Tuberculosis; Koch's Disease
Keywords: Atorvastatin; Anti-tuberculosis; HMG-COA Inhibitor; Statins; Anti TB drugs
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Atorvastatin; Isoniazid; Protons; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 20mg atorvastatin with standard of care (SOC) for TB (Experimental): Trial of 20mg atorvastatin with standard of care (SOC) for TB
  Interventions: Drug: Atorvastatin 20mg
- 40mg atorvastatin with standard of care (SOC) for TB (Experimental): Trial of 40mg atorvastatin with standard of care (SOC) for TB
  Interventions: Drug: Atorvastatin 40mg
- 60mg atorvastatin with standard of care (SOC) for TB (Experimental): Trial of 60mg atorvastatin with standard of care (SOC) for TB
  Interventions: Drug: Atorvastatin 60mg
- Standard of care (SOC) for TB (Active Comparator): Standard of care (SOC) for TB
  Interventions: Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamide (Z) Ethambutol (E)

INTERVENTIONS:
Drug: Atorvastatin 20mg — Participants will receive oral atorvastatin 20mg daily for 16 weeks
  Other Names: Astin
  Arms: 20mg atorvastatin with standard of care (SOC) for TB
Drug: Atorvastatin 40mg — Participants will receive oral atorvastatin 40mg daily for 16 weeks
  Other Names: Astin
  Arms: 40mg atorvastatin with standard of care (SOC) for TB
Drug: Atorvastatin 60mg — Participants will receive oral atorvastatin 60 mg daily for 16 weeks
  Other Names: Astin
  Arms: 60mg atorvastatin with standard of care (SOC) for TB
Drug: Fixed dose combination of Rifampicin (R) Isoniazid (H) Pyrazinamide (Z) Ethambutol (E) — Participants will receive 8 weeks of daily oral treatment with rifampin, isoniazid, pyrazinamide, ethambutol, followed by 16 weeks of daily oral treatment with rifampin, isoniazid
  Arms: Standard of care (SOC) for TB

SUMMARY:
Tuberculosis (TB) is caused by mycobacterial organism. It is the leading infectious disease cause of death globally. According to recent estimates from the World Health Organization (WHO), over 10 million new cases and 1.6 million deaths from TB occurred in 2021. The vast majority of TB cases and TB deaths are in developing countries. Nigeria has the highest TB burden in Africa with a high number of undetected TB cases as well. The spread of HIV has fueled the TB epidemic, and TB is the leading cause of death among patients infected with HIV and has assumed the lead position as the number one infectious disease cause of death globally. Even though the COVID-19 was associated with a huge mortality, TB contributed significantly to death and one of the single predictors of death among COVID-19 infected individuals. TB predominantly affects young adults in their most productive years of life and has substantial impact on economic development.

Emerging evidence has shown that lipid lowering drugs like statins can make the TB bacteria more susceptible to current treatment regimen. The ATORTUB group recently completed Phase II A and Phase IIB studies to assess the safety, tolerability and efficacy of atorvastatin when administered with the current standard of care. The investigators demonstrated that atorvastatin is well tolerated, save, and has beneficial microbiological and radiological impacts in tuberculosis, thus, warrants further studies.

This phase IIC trial sets out to evaluate the safety and efficacy of different doses of atorvastatin containing regimen, determine rate of decline of viable sputum bacilli, the time to stable sputum conversion, improvement in chest ray severity scores and lung function parameters post randomization in the different treatment arms. The phase II C is a Selection Trial with Extended follow-up STEP and has been devised as a pilot phase III where patients are studied for longer period (12months post randomization) than the usual phase IIB. Thus, providing additional data that will justify a successful phase III trial.

DETAILED DESCRIPTION:
INTRODUCTION Tuberculosis is a chronic disease responsible for most deaths from infectious disease with an estimated I0 million cases and close to 2 million deaths globally. Despite the availability of therapy for TB, the scourge of the disease has not abated especially in the developing countries. The disease is caused by a bacterium called Mycobacterium tuberculosis, a non-spore forming intracellular organism. TB exists in two forms; primary and secondary infection. While primary infection most times goes unnoticed and are usually associated with non-specific symptoms, secondary infections are usually associated with profound symptoms and signs in various organs especially in the lungs. Majority of persons overcome primary infection but the tubercule bacilli may lie dormant in the macrophages. Secondary infection occurs as a result of either endogenous reactivation or exogenous re-infection. Pulmonary TB is responsible for more than 85% of the cases.

MTB infect and survive humans by evading the various immune defense systems. The organism accumulates and utilizes an abundant amount of lipids and cholesterol for its cell wall, and as a source of carbon for synthesis of virulence factors. Mycobacterium tuberculosis also utilizes cholesterol as a vehicle to enter macrophage, inhibit phagocytosis and inhibit growth and development of phagocytes. These greatly impairs the hydrolytic and antimicrobial properties and activities of phagocytes. Current therapy is as old as the disease itself; is of long duration, hence it is associated with poor compliance. This contributes to frequent relapses and emergence of resistant form of the disease. Average interval between one episode of TB and another ranges from 6-18 months after completion of therapy. Despite clinical cure, approximately half of patients have permanent lung damage. In Nigeria, TB is a major risk factor for Chronic Obstructive Pulmonary Disease, lung fibrosis/scarring and other diseases. It is clear that new and innovative therapeutic agents are needed to tackle this hydra- headed disease. In order to address these challenges, a lipid lowering agent, atorvastatin is being repurposed.

The use of statins have been demonstrated in infectious diseases and especially in tuberculosis than other organisms. In vitro studies have demonstrated that statins could strengthen the host response against M. tuberculosis and inhibit the activation of T cells induced by M. tuberculosis antigens. In another study, murine bone marrow-derived macrophages that were exposed to simvastatin and were infected with M. tuberculosis, showed a significant reduction in mycobacterial growth, without adverse effects on cell viability. Treatment of TB in animal model with statins and anti TB drugs showed that treatment with anti-TB drugs plus simvastatin reduced the percentage of relapses by 50% compared with treatment with only anti-TB drugs. Taken together, all these studies in animal model indicate that statins has anti-TB effect, reduces bacillary load, shortens the duration of therapy and decreases relapse rate when used with first-line anti-TB drugs.

Most of the clinical evidence on the role of statins in TB were from retrospective and nested case control studies from Asian continent. In one study in Taiwan, diabetic subjects older than 65 treated with statins had a lower risk of developing active tuberculosis, with a risk of 0.76 (95% CI, 0.60-0.97). Chronic use of statins (more than 90 days) was associated with the lowest risk (RR 0.62; 95% CI 0.53-0.72) as shown in another study.

The ATORTUB investigators recently completed two phase 2 studies to assess the safety, tolerability and efficacy of atorvastatin administered with the current standard of care. The first study was a phase IIA study involving 40 patients randomized to receive standard of care alone and standard of care with oral (40mg) dose atorvastatin. Primary outcome at 2 weeks was safety, tolerability and early bactericidal activity over a 2 week period. The study showed that atorvastatin was generally safe and well tolerated. The rate of decline of colony forming unit was higher among the atorvastatin group. Even though there was no early bactericidal activity demonstrated at 2 weeks, atorvastatin group had significantly number of participants with more than 0.5 log10 decline in colony forming unit. This was quite significant. At the phase IIB study, 150 eligible participant's were randomly assigned to either of the two arms. All the participants had rifampicin sensitive active non complicated TB. Other drug resistance testing were not done. Oral dose of 40mg of atorvastatin was given for 2 months together with standard of care drugs and afterwards the standard of care drugs were continued for the patients to complete 6 months of therapy. Primary outcome were safety and tolerability atorvastatin , efficacy measured by the number of sputum conversion at 2 months. Secondary outcome was chest x-ray severity score at 2 months. AT the end of the phase IIB trial, it was shown that atorvastatin was generally safe and in fact participants in that group had reduced incidence of peripheral neuropathy. More participants achieved sputum conversion compared with the standard of care group. The mean improvement in chest x-ray severity score was higher in the experimental group Atorvastatin in combination with standard antituberculosis drugs achieved a significantly higher rate of sputum culture negativity and reduction in mycobacterial burden in sputum at 2 months compared with antituberculosis drugs alone. The difference in sputum negativity and the mean fall in colony forming unit per ml of sputum per month were significantly higher among the intervention group. The use of atorvastatin was also significantly associated with a negative sputum result. These may be indicative of the anti-mycobactericidal effect of atorvastatin, which had been earlier reported in murine models, other invitro studies and consistent with the earlier phase IIA result .

The ATORTUB investigators therefore concluded that atorvastatin has beneficial microbiological and radiological impacts in tuberculosis and warrants further studies.

Though, the phase IIB study reported positive findings that suggests the beneficial role of atorvastatin, however, before moving to a more expensive phase III study, important information relating to the clinical trial needs to be answered. For example, there is a need to establish the time to stable sputum conversion. This will be useful in determining the effective duration of atorvastatin containing regimen. In addition, evaluating the regimen among unbiased and diverse groups of patients including those with HIV, DM, hypertension and possibly children will be helpful and required. Even though, the dose we used was effective, conducting pk-pd evaluations at different doses and correlating these with outcomes of the trial will be essential.

Phase IIC also referred to as Selection Trial with Extended follow-up STEP, has been devised as a pilot phase III where patients are studied for longer period than the usual phase IIB and additional data that will justify and ensure a successful phase III trial are obtained. Patients are followed up for a fairly longer time in phase IIC , 12 months post randomization.

2. Study Design

Experimental design/Research Plan This is a multicenter, randomized, controlled, open-label, 4-arm, phase IIC superiority trial.

For the phase III aspect, the study will be fully international and multicenter.

Phase IIC will seek to determine the safety and efficacy of different doses of atorvastatin containing regimen , the time to sputum culture conversion, time to decline in Chest x-ray severity score and improvement in lung function parameters by atorvastatin at mentioned doses in combination with standard anti-TB regimen in 440 patients.

Consented and eligible patients aged12 -65 years with active tuberculosis will be recruited and have study-specific procedures initiated at enrollment / Screening visit. At screening visit, participants will be interviewed for demographics, contact information, medical history. They will have their anthropometry documented, will be screened for HIV, Diabetes and Pregnancy (in females), and have sputum collected for mycobacterial smear and culture.

At baseline visit (visit at which study drug is initiated), sputum will be collected for mycobacterial smear and culture, blood sample for complete blood count, serum or plasma for alanine aminotransferase (ALT), total bilirubin, creatinine, albumin, and potassium, complete lipid profile, creatine phosphokinase, unless results from those tests performed within fourteen days prior to screening are available. Sweat test and lung function test will be performed prior randomization. In this visit (baseline), participants will be randomized to receive either 20/40/60mg of daily treatment with atorvastatin for 16 weeks (from the beginning of standard of care treatment) with standard anti-TB regimen (2RHZE/4RH) for 24weeks (6 months) or the standards anti-TB drugs alone for 24 weeks (6 months). Randomization will be stratified by site, by HIV status (HIV-uninfected vs. HIV- infected with CD4 T cell count greater than or equal to 200 cells/mm3 vs. HIV-infected with CD4 T cell count less than 200 cells/mm3) and by DM status (DM patients vs. non-DM) and will follow a predefined allocation ratio of 1:1:1:1. Thereafter, participants will be followed up closely up to 12 months post randomization (i.e. study specific procedures will be carried out at weeks 2,4,6,8,10,12, 16, 22, 24; months 8, 10 and 12 post randomization according to study protocol). During this period, the number and types of Adverse Events in the participants will also be reported and documented.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all the following inclusion criteria in order to participate in this study:

A. Suspected pulmonary tuberculosis plus one or both of the following: a) at least one sputum specimen positive for acid-fast bacilli on smear microscopy OR b) at least one sputum specimen positive for M. tuberculosis by Xpert MTB/RIF testing, with semiquantitative result of 'medium' or 'high' and rifampicin resistance not detected.

B. Treatment naive

C. Age twelve years or older

D. A verifiable address or residence location that is readily accessible for visiting, and willingness to inform the study team of any change of address during the treatment and follow-up period.

E. Documented HIV infection status.

F. Documented blood sugar level/ Diabetes

G. For HIV-positive individuals, CD4 T cell count greater than or equal to 100 cells/mm3 based on testing performed at or within 30 days prior to screening.

H. Laboratory parameters done at or within 14 days prior to screening:

* Serum or plasma alanine aminotransferase (ALT) less than or equal to 3 times the upper limit of normal
* Serum or plasma total bilirubin less than or equal to 2.5 times the upper limit of normal
* Serum or plasma creatinine level less than or equal to 2 times the upper limit of normal
* Serum or plasma potassium level greater than or equal to 3.5 meq/L
* Hemoglobin level of 7.0 g/dL or greater
* Platelet count of 100,000/mm3 or greater

I. For women of childbearing potential, a negative pregnancy test at or within seven (7) days prior to screening

J. Written informed consent

Exclusion Criteria:

Individuals with any of the following exclusion criteria at the time of enrollment or initiation of study drugs will be excluded.

A. Pregnant or breast-feeding

B. Unable to take oral medications

C. Those already on treatment for tuberculosis

D. Weight less than 40.0 kg

E. Known allergy or intolerance to any of the study medications

F. Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any one or more of the following: rifampin, isoniazid, pyrazinamide,or ethambutol,

G. .Evidence of clinically significant metabolic or co morbid medical conditions ; malignancy; or other diseases like history of or current cardiovascular disorder such as heart failure, coronary heart disease, arrhythmia.

H. Known or family history of bleeding disorders. I. Any renal impairment characterized by serum creatinine clearance of 1.5 x upper limit of normal of the clinical laboratory reference range at screening.

J. Myositis and or Creatinine phosphokinase three times upper limit of normal K. Other medical conditions, that, in the investigator's judgment, make study participation not in the individual's best interest.

Criteria for Exclusion after Enrollment ('Late Exclusion')

Microbiological confirmation of drug-susceptible tuberculosis is not expected always to be available at the time of enrollment. Enrolled individuals who are subsequently determined to meet either of the following criteria will be classified as 'late exclusions' and study treatment will be discontinued:

A. Screening, baseline, and Week 2 study visit sputum cultures all fail to grow M. tuberculosis.

B. M. tuberculosis cultured or detected through molecular assays (Cepheid Xpert MTB/RIF or Hain MTBDRplus assays) from sputum obtained around the time of study entry is determined to be resistant to one or more of isoniazid, rifampin, or fluoroquinolones.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Proportion of participants with grade 3 or higher adverse events during study drug treatment | for 24 weeks post randomization
  Proportion of participants with grade 3 or higher adverse effect as measured by (CTCAE) v5.0
Efficacy: TB disease-free survival at six months post randomization | six months post randomization
  The proportion of participants with TB disease-free survival post randomization
  * They have negative sputum culture.
  * if at the end of the follow-up period, they are clinically without symptoms/signs of ongoing active TB and are unable to produce a sputum specimen
  * If at the end of the follow-up period they are clinically without symptoms/signs of ongoing active TB and produce a sputum without evidence of M. tuberculosis
  * if at the end of the follow-up period, they have at least 30% improvement in chest severity score and 15% improvement in spirometric values.
Efficacy:Time to stable sputum culture conversion on solid and /liquid media | up to 24 weeks post randomization
  Time to achieve culture negative sputum result as measured by growth on solid mycobacteria culture medum
Efficacy: Proportion of participants who are culture negative | Up till 24 weeks post randomization.
  Proportion of participants who have Sputum culture negative specimens at the end of treatment

SECONDARY OUTCOMES:
Efficacy: TB disease-free survival at twelve months post randomization | 52 weeks post randomization
  Proportion of participants with no TB disease
Efficacy: Proportion of participants who are symptom free at 12 months post randomization | 52 weeks post randomization
  Proportion of participants who are symptom free at 12 months post randomization will be presented as frequency.
Efficacy: Proportion of participants with improved chest x-ray severity | 52 weeks post randomization
  Proportion of participants with at least 30% reduction in Chest x-ray severity as measured by Timika score
Efficacy: Proportion of participants with improvement in lung function post treatment | Up till 52 weeks post randomization.
  Proportion of participants with at least 15% improvement in FEV1 and FVC post measured by Spirometry

OTHER OUTCOMES:
Diagnostic utility of Sweat TB test | At enrolment
  Sensitivity and specificity of Sweat TB test in comparision with TB culture

CONTACTS AND LOCATIONS:
Overall Officials: Olanisun O Adewole, MD, Principal Investigator — Obafemi Awolowo University /Teaching Hospital, Ile- Ife, Osun State, Nigeria; Olanisun O Adewole, MD, Study Chair — Obafemi Awolowo University/ Teaching Hospital, Ile- Ife, Osun State, Nigeria; Bolanle A Omotoso, MD, Study Director — Obafemi Awolowo University/ Teaching Hospital, Ile- Ife, Osun State, Nigeria
Locations (8):
- Nigeria (8):
  - National Tuberculosis Reference Laboratory, Zaria, Kaduna State
  - Federal Teaching Hospital, Katsina, Katsina State
  - Federal Medical Center, Keffi, Nasarawa State
  - Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Osun State
  - Bowen University Teaching Hospital, Iwo, Osun State
  - University College Hospital, Ibadan, Oyo State
  - Usman Danfodio University, Sokoto, Sokoto State
  - University of Abuja Teaching Hospital, Gwagwalada

IPD SHARING:
Plan to Share IPD: No